CLINICAL TRIAL: NCT03041714
Title: Neurophysiologic Study of Patients With Essential Tremor and Dystonic Tremor
Brief Title: Neurophysiologic Study of Patient With Essential Tremor and Dystonic Tremor
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170053; 17-N-0053
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-03

CONDITIONS: Essential Tremor; Cervical Dystonia; Focal Dystonia
Keywords: Essential Tremor; Cervical Dystonia; Hand Dystonia; Neurophysiology; Dystonic Tremor
MeSH Terms: conditions — Essential Tremor; Torticollis; Dystonic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Normal volunteers: people who are healthy and without tremor
- Essential tremor: Patients with essential tremor
- Dystonic tremor: patient with tremor who also have dystonia

SUMMARY:
Background:

Essential tremor is when a person has tremor, but no other neurological symptoms. Dystonic tremor is when a person also has dystonia. Dystonia is a condition in which muscle contraction causes changes in posture. Researchers do not fully know what areas of the brain cause these tremors, or how the types differ. They also do not know what tests can identify the differences.

Objective:

To look at differences between essential tremor and dystonic tremor.

Eligibility:

People ages 18 and older with or without tremor

Design:

Participants will be screened with medical history, physical exam, and urine tests. Those with tremor will complete questionnaires about how tremor affects them.

The screening and study visits can be done on the same day or on separate days.

Participants will have 1 or 2 study visits. These include magnetic resonance imaging (MRI) and tremor testing.

For MRI, participants will lie on a table that slides in and out of a cylinder that takes pictures. Sensors on the skin measure breathing, heart rate, and muscle activity. This takes about 2 hours.

Tremor testing will include transcranial magnetic stimulation (TMS), electrical stimulation of the fingers, doing a movement task, and recording of tremor movements. For TMS, two wire coils will be held on the scalp and a brief magnetic field will be produced. A brief electrical current will pass through the coils. For the other tests, small sticky pad electrodes will be put on the skin. Participants will move their hand when they hear a sound. They will get weak electrical shocks to their fingers. These tests will take 3-4 hours.

Participants can take part in either or both parts of the study.

DETAILED DESCRIPTION:
Objectives:

To explore a neurophysiological difference between patients with essential tremor (ET) and dystonic tremor (DT).

Sample Size and Population:

We plan to recruit 26 healthy volunteers (HVs), 26 patients with ET, 26 patients with dystonic tremor from the Movement Disorders and Botulinum Toxin (BoNT) clinics of HMCS. The dystonic tremor group will be divided into 2 subgroups: pure dystonic tremor (pDT), patients who have dystonia and tremor in the same limb, tremor associated with dystonia (TAWD), patients who have isolated tremor with dystonia elsewhere. We plan to enroll 13 patients with pDT and 13 with TAWD. We plan to recruit a total of 20 participants including patients with ET, DT and HVs if the use of data from protocol 10-N-0009 is permitted. All neurophysiologic results will be compared between patients and HVs.

Design:

Subjects will come to NIH for at least one study visit. All subjects will undergo a screening visit including taking a medical history and physical examination. Then the patients will be scored clinically for tremor in both ET and DT and dystonia only for DT. All subjects will have a series of transcranial magnetic stimulation (TMS) studies. TMS-induced electromyographic (EMG) activity of hand and forearm muscles will be recorded as motor evoked potentials (MEPs). Pyramidal threshold will be determined by inion stimulation. Then, paired-pulse stimulation at the cerebellum followed by the motor cortex will be performed at rest and at tonic activation of the hand muscle. Only patients will have recordings of tremor at rest, postural holding, and with action and specific tasks such as writing by using accelerometry and EMG. Additionally, a single TMS will be delivered to the motor cortex or cerebellum while the patients elicit their tremor in order to explore the effect of TMS on tremor. All subjects (both HVs and ET, DT) will be tested for their threshold to discriminate somatosensory stimulation and for their performance of quick ballistic movements. All subjects will also undergo a magnetic resonance imaging (MRI) study which includes structural MRI, resting state functional MRI (rsfMRI), diffusion tensor imaging (DTI), MR spectroscopy. The subjects can either undergo the MRI study on the same visit as the other parts of experiment or do it separately.

Outcome measurements:

The various neurophysiological results include the data from the TMS experiment, tremor analysis, threshold of temporal discrimination, ballistic movement and MRI experiment. These results will be compared between HVs and patients group.

ELIGIBILITY:
* INCLUSION CRITERIA

Tremor Subjects:

* Must be 18 years or older
* Fulfill the diagnostic criteria of essential tremor, pure dystonic tremor and tremor associated dystonia, as defined by the Consensus Statement of the Movement Disorder Society on Tremor, 1998. We will recruit patients displaying hand tremors in each group as the follows:

  * Hand tremor patients in ET group.
  * Dystonic hand tremor patients in pDT group.
  * Cervical dystonia (CD) patients or spasmodic dysphonia and hand tremor without clinical evidence of hand dystonia in TAWD group.
* Ability to give informed consent.
* Ability to comply with all study procedures, based on the judgment by the investigator(s).
* Agree to not drink caffeine or alcohol for 48 hours before participating in the protocol.

Healthy Volunteers:

* Must be 18 years or older
* Absence of dystonia or other neurological disorder with any effect on the motor or sensory systems.
* Ability to give informed consent.
* Ability to comply with all study procedures, based on the judgment by the investigator(s).
* Agree to not drink caffeine or alcohol for 48 hours before participating in the protocol.

EXCLUSION CRITERIA:

Patients:

* Botulinum toxin treatment < 3 months prior to visit.
* Employees and/or staff of NINDS
* Has used illegal drugs within the past 6 months based on history. The intent is to exclude those with drug use that may affect study results. Participants who appear to be intoxicated at the time of testing will be rescheduled.
* Has more than 7 alcoholic drinks a week in the case of a woman and 14 alcoholic drinks a week in the case of a man.
* Abnormal findings on neurologic exam (other than tremor and dystonia in patient group)
* Has had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures.
* Has major depression or any major mental disorders (axis I disorders)
* Has a neurologic disorder other than tremor or dystonia
* Has had a head injury where there was a loss of consciousness for more than a few seconds.
* Currently taking primidone, anticholinergics or benzodiazepines.

Healthy Volunteers:

* Employees and/or staff of NINDS
* Has used illegal drugs within the past 6 months based on history. The intent is to exclude those with drug use that may affect study results. Participants who appear to be intoxicated at the time of testing will be rescheduled.
* Has more than 7 alcoholic drinks a week in the case of a woman and 14 alcoholic drinks a week in the case of a man.
* Abnormal findings on neurologic exam.
* Has had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures.
* Has a neurologic disorder other than tremor or dystonia
* Has major depression or any major mental disorders (axis I disorders)
* Has had a head injury where there was a loss of consciousness for more than a few seconds.

Additional Exclusion Criteria for MRI:

* Has metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, or metal fragments in the eye
* Pregnancy
* Unable to lie flat on the back for the expect length of the study up to 3 hours.
* Feeling uncomfortable being in a small space for up to 3 hours.

<TAB>

Additional Exclusion Criteria for TMS:

* Has metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, or metal fragments in the eye
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be referred to NIH or may refer themselves from all over the United States.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
The various neurophysiological results including the data from TMS experiment, tremor analysis, threshold of temporal discrimination, ballistic movement and MRI experiment. These results will be compared between HVs and patients group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Deuschl G, Bain P, Brin M. Consensus statement of the Movement Disorder Society on Tremor. Ad Hoc Scientific Committee. Mov Disord. 1998;13 Suppl 3:2-23. doi: 10.1002/mds.870131303. PMID 9827589
- [Background] Ni Z, Pinto AD, Lang AE, Chen R. Involvement of the cerebellothalamocortical pathway in Parkinson disease. Ann Neurol. 2010 Dec;68(6):816-24. doi: 10.1002/ana.22221. PMID 21194152
- [Background] Pascual-Leone A, Valls-Sole J, Toro C, Wassermann EM, Hallett M. Resetting of essential tremor and postural tremor in Parkinson's disease with transcranial magnetic stimulation. Muscle Nerve. 1994 Jul;17(7):800-7. doi: 10.1002/mus.880170716. PMID 8008009